CLINICAL TRIAL: NCT05407662
Title: REal-world Use of steroidaL mIneralocorticoid reCeptor Antagonists - the RELICS Study - Patient Survey (PS)
Brief Title: A Study Using Surveys to Learn More About Treatment With Steroidal Mineralocorticoid Receptor Antagonists, How They Are Used, What Side Effects They Have, and How Satisfied People Who Receive Them Are in the US
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 22114
Record Dates: First submitted 2022-06-02; First posted 2022-06-07 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Chronic Kidney Disease; Type 2 Diabetes Mellitus; Heart Failure
MeSH Terms: conditions — Renal Insufficiency, Chronic; Diabetes Mellitus, Type 2; Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

GROUPS / COHORTS (1):
- Survey on users of sMRA therapies: sMRA stands for steroidal mineralocorticoid receptor antagonist.
  Interventions: Other: sMRA therapies

INTERVENTIONS:
Other: sMRA therapies — No drug will be provided to participants. Patients follow routine clinical practice/administration.
  Other Names: Steroidal mineralocorticoid receptor antagonist therapies

SUMMARY:
This is an observational study in which patients with chronic kidney diseases (CKD), type 2 diabetes (T2D) or heart failure (HF) who are current or past users of sMRA therapies are studied. sMRA stands for steroidal mineralocorticoid receptor antagonists.

CKD is a long-term, progressive decrease in the kidneys' ability to work properly.

Type 2 diabetes is a condition in which the body does not make enough of a hormone called insulin or does not use insulin well resulting in high blood sugar levels.

HF is a condition in which the heart does not pump blood as well as it should.

The renin-angiotensin-aldosterone system (RAAS) is a hormone system that works with the kidneys to control blood pressure and the balance of fluid and electrolytes (like salt) in the blood. The RAAS has been a treatment target of heart and kidney diseases for decades. One of these classes of medications is called mineralocorticoid receptor (MR) antagonists (MRAs). MRAs work to directly block the action of a hormone called aldosterone. Aldosterone is produced naturally by the adrenal glands, and it can increase the blood volume and blood pressure. Using MRAs therapies can help prevent strokes, heart attacks and kidney problems.

Spironolactone was the first available MRA in the US with its approval in 1960. Eplerenone is another MRA which has been available since 2002. Both spironolactone and eplerenone are known as steroidal MRA (sMRA) due to their chemical structures.

The main purpose of this study is to collect more data on the characteristics of patients who are taking sMRA currently and those who have discontinued sMRA therapy in the past 12 months.

To do this, patients who have received sMRA in the most recent 12 months will be invited to participate in the study and asked to complete surveys if they agree to join the study. Patients will be found from administrative claims in a database called HealthCore Integrated Research Database (HIRD).

And the other purposes of the study are to learn more about:

* the indications for sMRA therapy
* the frequency and symptoms of reported side effects of sMRA treatment
* the treatment satisfaction and effectiveness as well as potential reasons for treatment continuation/discontinuation of sMRA therapies

Besides this data collection, no further tests or examinations are planned in this study.

The participants will receive their treatments as prescribed by their doctors during routine practice according to the approved product information.

Researchers will look at the health information from adult men and women in the US only if applicable who are current/past users of sMRA therapies with diagnosis of CKD or T2D or HF, consent to participate in the study.

ELIGIBILITY:
Inclusion Criteria:

* Currently active with commercial or Medicare Advantage health insurance (both medical and pharmacy benefits) at the time the patient sample is identified
* ≥1 pharmacy claim for a sMRA therapy (spironolactone or eplerenone) in the most recent 12-months of claims data
* ≥1 inpatient or ≥2 outpatient medical claims with an International Classification of Diseases, Ninth/Tenth Revision, Clinical Modification (ICD-9/10-CM) diagnosis code for CKD, T2D or HF going back to 1 Jan 2006
* Age ≥18 years at the end of the patient identification period
* Has email and/or mailing address
* Consent to participate in the survey

Exclusion Criteria:

- None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are current/past users of sMRA therapies who were diagnosed with chronic kidney disease, type 2 diabetes mellitus or heart failure, consent to participate in the study and have a valid survey.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Actual)
Dates: Start 2022-11-02 (Actual); Primary Completion 2023-06-13 (Actual); Study Completion 2023-06-13 (Actual)

PRIMARY OUTCOMES:
Screening questions - to verify the participant's basic information and current health plan status and validate their current or recent use of sMRA therapy | Up to 12 months
  sMRA stands for steroidal mineralocorticoid receptor antagonists.
Condition history - to confirm the diagnosis of CKD, T2D, or HF, determine the age at condition diagnosis, and the type of physician who currently manages/treats condition | Up to 12 months
sMRA discontinuer questions - questions for patients who have discontinued sMRA therapies, including duration of use, how long ago discontinued and most recent dose | Up to 12 months
sMRA continuing user questions - questions for patients who are current sMRA users including current sMRA therapy, how long used and most recent dose | Up to 12 months
Clinical characteristics | Up to 12 months
Demographic characteristics | Up to 12 months
Claims-based patient characteristics | Up to 12 months
Baseline comorbid conditions of interest | Up to 12 months
Baseline sMRA adherence and persistence | Up to 12 months
Baseline all-cause healthcare resource utilization by place of service | Up to 12 months
Baseline all-cause healthcare costs by place of service | Up to 12 months

SECONDARY OUTCOMES:
sMRA discontinuer questions - targeted past medical history (indications for sMRA therapy) , reasons for choosing/discontinuing to sMRA therapy | Up to 12 months
sMRA continuing user questions - targeted past medical history (indications for sMRA therapy), reasons for choosing/continuing to use current sMRA | Up to 12 months
sMRA discontinuer questions - occurrence of sMRA side effects | Up to 12 months
sMRA continuing user questions - occurrence of sMRA side effects | Up to 12 months
sMRA discontinuer questions - reasons for discontinuing sMRA therapy, perceived effectiveness and overall satisfaction with the sMRA therapy | Up to 12 months
sMRA continuing user questions - Treatment Satisfaction Questionnaire for Medication version 1.4 (TSQM v1.4) - validated PROM the evaluates patients' perception of sMRA treatment effectiveness, convenience, and overall satisfaction | Up to 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Many Locations, Whippany, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.